CLINICAL TRIAL: NCT01115400
Title: Quality of Life Evaluations in Patients With Abdominal Wall Hernias
Acronym: QOL
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-07-31; 05-07-31 (Other: University Hospitals Case Medical Center)
Record Dates: First submitted 2010-04-12; First posted 2010-05-04 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Hernia
Keywords: Abdominal Wall Hernia; quality of life
MeSH Terms: conditions — Hernia; Hernia, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. The investigators would like to use this survey to elucidate how quality of life of the patient is changed with the presence of an abdominal wall hernia.

DETAILED DESCRIPTION:
Abdominal hernia repair is one of the most common general surgery procedures performed in the United States. Hernia occurrences after prior abdominal surgeries can range anywhere from 20-50%. Small abdominal defects (<3cm) can generally be repaired primarily, however, anything larger usually requires placement of mesh. If the defects are massive and complicated from prior repairs; they often require prolonged operating time, and sometimes even multiple-staged procedures to complete repair. In patients with co-morbidities and needing abdominal hernia repair, the surgeons are generally cautious in recommending surgical treatments as long as no acute emergency exists due to the hernia. Due to the high post-operative complications in these patients, the risks of the surgery may outweigh the benefit of the repair. As a result, many patients with large, complicated hernias are delegated to medical management including the use of abdominal binders, conservative treatments of enterocutaneous fistula and chronic infections. However, these decisions are frequently made from the point of the view of the surgeons, and not the patients.

The investigators would like to evaluate how the patients perceive living with abdominal hernias, and how they view the effect of their quality of life affected by hernias. If the quality of life in these patients is severely affected, the investigators may be able to use that information to stratify these patients and to gauge the necessity of future repairs.

Currently, there is no quality of life survey target specifically for patients with abdominal hernia. Most institutions use the SF36 or a shortened SF36 form to evaluate quality of life. However, the SF36 is generic and cumbersome. It was originally designed for renal failure patients and is not entirely appropriate for hernia patients. This protocol will be the first one to use factors that are specific to hernia patients to accurately describe the patient's quality of life. Also, by generating a quality of life score for patients with different degrees of hernias, the investigators will be able to better stratify patients who may benefit from the hernia repair more than what the surgeons perceive because of the patients' other co-morbidities. And furthermore, the investigators would also like to show the improvement in quality of life in these patients after their successful repairs.

The Hernia QOL survey will be compared with the SF12 (a shortened version of the SF36).

ELIGIBILITY:
Inclusion criteria:

* Subjects who are 18 years of age and older
* Subjects of either sex
* Subjects with the diagnosis of abdominal wall hernias
* Subjects who agree to participate in the study program

Exclusion criteria:

* Subjects who present to clinic with acute incarceration or strangulation of bowel
* Subjects who are unable to read or write to complete the survey
* Pregnant women, minors, psychiatric patients and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This protocol will involve patients presenting to University Hospitals Case Medical Center for evaluation of abdominal hernias.
  The study population will include all adult patients with the diagnosis of abdominal wall hernias, without incarceration or strangulation of bowels. The investigators will need about 90 subjects to participate in this study.
  The survey will be entirely anonymous; no patient information will be given out in any part of the survey.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Quality of life perception | up to 1 year
  The investigators would like to evaluate how the patients perceive living with abdominal hernias, and how they view the changes from their baseline in their quality of life since their hernia. If the quality of life in these patients is severely affected,the investigators may be able to use that information to stratify these patients and to gauge the necessity of future repairs

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rosen, MD, Principal Investigator — Univesity Hospitals Case Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States